CLINICAL TRIAL: NCT00314522
Title: Optimization of Spectroscopic Imaging Parameters and Procedures for Prostate at 3 Tesla Using an External Probe
Status: Completed | Type: Observational
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Cross Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: EX-0003
Record Dates: First submitted 2006-04-11; First posted 2006-04-14 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2011-12

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

SUMMARY:
This study performed a retrospective analysis of patient images to develop software in determining dose delivered for each fraction treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subject 18 years of age and over

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clniic
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2005-09; Study Completion 2006-03

CONTACTS AND LOCATIONS:
Overall Officials: Gino Fallone, PhD, Principal Investigator — AHS Cancer Control Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada